CLINICAL TRIAL: NCT02560090
Title: Transforming Patient-Centered Medical Homes Into Medical Communities for Underserved Rural Patients
Brief Title: Bamberg Diabetes Transitional Care Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); South Carolina Department of Health and Human Services (Unknown); North Carolina Translational and Clinical Sciences Institute (Other); The Regional Medical Center of Orangeburg and Calhoun Counties (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00038334
Record Dates: First submitted 2015-07-15; First posted 2015-09-25 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Survey assessments as well as collection of medical records and billing information.
  Interventions: Behavioral: Surveys
- Telephonic Nurse Intervention (Active Comparator): Survey assessments as well as collection of medical records and billing information. A nurse will communicate with participants via telephone to support diabetes self-management practices.
  Interventions: Behavioral: Surveys; Behavioral: Telephonic Nurse Intervention
- In-person Community Health Worker Intervention (Active Comparator): Survey assessments as well as collection of medical records and billing information. A community health worker will work with participants in person to support diabetes self-management practices.
  Interventions: Behavioral: Surveys; Behavioral: In-person Community Health Worker

INTERVENTIONS:
Behavioral: Surveys — The following information will be collected: demographics, literacy screener, depression screener, medication adherence, self-efficacy, tobacco use, patient activation, health questionnaire, eating patterns, diabetes self-management assessment, stages of change questionnaire, vitals, and self-care behaviors.
Behavioral: Telephonic Nurse Intervention — A nurse will contact patients by phone at least weekly for month 1 and at least every other week for months 2 and 3 and will collect the following information: medication adherence, discharge plan adherence, problem solving, diet and physical activity issues and to assess self-management, dietary, and physical activity improvements. In addition the nurse will link participants with resources.
  Arms: Telephonic Nurse Intervention
Behavioral: In-person Community Health Worker — An in-person Community Health Worker will contact patients in-person at least weekly for month 1 and at least every other week for months 2 and 3 and will collect the following information: medication adherence, discharge plan adherence, problem solving, diet and physical activity issues and to assess self-management, dietary, and physical activity improvements. In addition the nurse will link participants with resources.
  Arms: In-person Community Health Worker Intervention

SUMMARY:
Bamberg County residents who has been diagnosed with or is at high risk for diabetes, may be eligible for a clinical research study to improve diabetes self-management and decrease hospital re-admissions.

The purpose of this study is to compare the effectiveness of three hospital discharge follow-up methods:

1. standard of care,
2. a nurse telephone intervention (care coordination and education), and
3. an in-home community health worker intervention (care coordination and education).

ELIGIBILITY:
Inclusion Criteria:

* Bamberg County resident
* between 18 and 75 years of age
* a patient discharged from the Regional Medical Center emergency department or Regional Medical Center hospital within 72 hours prior to consent
* diagnosed with diabetes or at high risk for diabetes
* will be a Regional Medical Center patient for follow-up care
* speaks English
* has access to a phone

Stage 2 Recruitment:

* If recruitment at 3 weeks after the first patient is enrolled is < 15 or the recruitment at 12 weeks is < 45, additional inclusion criteria will include the following: Regional Medical Center outpatient or unassigned community member with uncontrolled diabetes (defined as A1C >8 or blood pressure >140/90) is uninsured or who self-reports problems with obtaining medications.

Exclusion Criteria:

* end-stage renal disease
* terminal illness (e.g., advanced cancer, end-stage chronic obstructive pulmonary disease, advanced dementia)
* incarceration
* resident in a skilled nursing home.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change of Number of Hospital Re-admissions from 2 Years Prior to Study Enrollment to 1 Year After Study Completion | Retrospective billing collection 2 years prior to study enrollment and 1 year after study completion
  Hospital data will be obtained from Revenue and Financial Affairs South Carolina Data Oversight Council. These data come from the health organization where patients receive care and include components such as age, health care facility type, dates of admission/ discharge, length of stay, charges, payment source, primary and secondary procedure codes.
Change of Self-management Success Measured by Diabetes Self-Management Assessment Survey Tool from Baseline to Study Completion | Baseline, 1 month post-enrollment, 2 months post-enrollment, 3 months post-enrollment (study completion)
  Diabetes self-management assessment tool administered to participant over the phone or in-person

SECONDARY OUTCOMES:
Change of Health Goal Progress Captured by Field Notes to Track Intervention Activities from Baseline to Study Completion | Baseline, 1 month post-enrollment, 2 months post-enrollment, 3 months post-enrollment (study completion)
  Field Notes are completed after each interventionist's interaction with the participant to track progress to addressing health goals
Change of Diet Measured By a 24-item Introduction to the Lifestyle Survey from Baseline to Study Completion | Baseline, 1 month post-enrollment, 2 months post-enrollment, 3 months post-enrollment (study completion)
  The 24-item Introduction to the Lifestyle Survey will be used to assess diet (fats, protein, fruits and vegetables) and at enrollment, week 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Jenkins, DrPh, MSN, Principal Investigator — Medical University of South Carolina; Samuel Cykert, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The Regional Medical Center of Orangeburg and Calhoun Counties, Orangeburg, South Carolina, United States